CLINICAL TRIAL: NCT03869112
Title: The Effectiveness of a Physical Activity Intervention Versus Pulmonary Rehabilitation on Cardiovascular Risk Markers for Individuals With Chronic Obstructive Pulmonary Disease: a Feasibility Study
Brief Title: Physical Activity Intervention and Cardiovascular Risk Markers in COPD
Acronym: PARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Loughborough University (Other)
Responsible Party: Principal Investigator, Tareq Alotaibi, Principal investigator, University Hospitals, Leicester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18/EM/0270
Record Dates: First submitted 2019-02-26; First posted 2019-03-11 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; COPD
Keywords: COPD; Physical activity; pulmonary rehabilitation; COPD physical activity level; COPD comorbidities
MeSH Terms: conditions — Cardiovascular Diseases; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: A feasibility study with three groups. two interventional groups and one control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical activity intervention (Experimental): Physical activity group will be given a FitBit device to monitor their PA, especially steps count Step targets will be discussed with the participants with a view to increasing their daily physical activity over the 6 week period. A recent protocol has been described that encouraged an increase of 500 steps weekly. This was well tolerated by participants (Demeyer, Louvaris et al. 2017). This will be an unsupervised, home based intervention.
  Interventions: Behavioral: Physical activity intervention
- Pulmonary rehabilitation group (Experimental): Pulmonary rehabilitation group is a 6-week intervention of supervised exercise and group education and will follow the BTS guidelines. (Bolton, Bevan-Smith et al. 2013)
  Interventions: Other: Pulmonary rehabilitation group
- Usual care (No Intervention): Usual care group will have the standard follow up care by rehabilitation clinic without being in any physical intervention.

INTERVENTIONS:
Behavioral: Physical activity intervention — Physical activity group will be given a charge 2 FitBit device to monitor their PA specially steps count, step targets will be discussed with the participants with a view to increasing their daily physical activity over the 6 week period. A recent protocol has been described that encouraged an increase of 500 steps weekly. This was well tolerated by participants (Demeyer, Louvaris et al. 2017). This will be an unsupervised, home-based intervention.
  Arms: Physical activity intervention
Other: Pulmonary rehabilitation group — Pulmonary rehabilitation group is a 6-week intervention of supervised exercise and group education and will follow the BTS guidelines. (Bolton, Bevan-Smith et al. 2013)
  Other Names: Exercise intervention
  Arms: Pulmonary rehabilitation group

SUMMARY:
The Aim of this study is to examine the feasibility of a future trial comparing the impact of a physical activity intervention and a standard pulmonary rehabilitation programme upon cardiovascular risk and symptoms in COPD. The study involved three groups which are physical activity group, pulmonary rehabilitation group and usual care. The physical activity group and the pulmonary rehabilitation group will complete six-weeks of intervention. The pulmonary rehabilitation group will participate in a standard rehabilitation programme of supervised exercise and education sessions. Physical activity group will be involved in a programme that aims to increase their physical activity level with an increasing step count. Usual care group will be monitored for six-weeks.

Before and after interventions measures will be taken including exercise capacity, body composition, blood tests, arterial stiffness, questionnaires assessing health quality of life, anxiety and depression, symptoms, cardiovascular disease risk.

The investigators will also have a sub-group study. The subgroup study will have two arms interventions which are pulmonary rehabilitation group and physical activity group. The investigators will recruit 10 participants for each group from the main groups' population (no usual care group). Additional before and after measures will be taken for sub-group study and that includes Magnetic resonance imaging (MRI) scanning for adipose visceral tissue and postprandial lipaemic response test.

It is hypothesised that exercise and physical activity level can reduce cardiovascular disease risk with COPD patients, but the relative impact of both interventions need to be explored.

DETAILED DESCRIPTION:
For those with COPD, both physical activity (PA) interventions and pulmonary rehabilitation (PR) seem to be promising to potentially lower the risk of CVD. PA interventions seem to be promising in improving outcomes of COPD but there is lack of evidence on how the effectiveness of PA interventions compared with the gold standard intervention of PR.

However, the outcomes of both interventions have not been extensively investigated, nor have they been directly compared. The immediate effects of pulmonary rehabilitation and PA interventions on cardiovascular risk factors for individuals with COPD have not been extensively investigated or compared.

Therefore, the purpose of this study is to examine the feasibility of conducting a trial to compare the impact of pulmonary rehabilitation and physical activity interventions in a number of important clinical outcomes including cardiovascular risk.

Investigation and data collection will be taking place within University Hospitals of Leicester NHS trust sites. The investigators are aiming to recruit 50 COPD patients who are eligible for a pulmonary rehabilitation programme to investigate the effect of physical activity intervention compared to pulmonary rehabilitation with respect to cardiovascular risks.

The study will measure various outcomes, immediately before, immediately after interventions. These outcomes will include measures in aerobic fitness (walking test), strength tests, physical activity level, quality of life, breathlessness questionnaires. In addition, blood sampling and body measurements will be completed. The investigators will also measure arterial stiffness with a non-invasive technique. Arterial stiffness is a hardening of the artery wall.

In a subgroup study, 20 participants will have additional visits and measures. The investigators will be doing magnetic resonance imaging (MRI), diagnostic pictures of the inside of the body which is used for picturing the fat tissue around the abdomen. The investigators will be also doing a postprandial lipaemic test which is testing the fat level in the circulating blood after a high-fat meal. The investigators will do this test as before and after the intervention to allow for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 40 years to 85 years.
* Diagnosed with COPD
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Participant is willing to attend visits at baseline and 8 weeks (sub-group: baseline, 8 weeks)
* Able to read and understand English

Exclusion Criteria:

* Age <40
* Attended a pulmonary rehabilitation programme or participating in a physical activity intervention study in current time or in the last 6 months.
* Any other significant diseases or disorders that are a contraindication to be enrolled in a pulmonary rehabilitation programme.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | Change from baseline waist circumference at 8 weeks.
  Waist circumference will be determined at the narrowest part of the torso above the umbilicus and below the xiphoid process using a measuring tape before and after the intervention.
Body fat percentage | Change from baseline body fat percentage at 8 weeks.
  Body fat in percentage will be measured in %BF using bioelectrical impedance analysis before and after the intervention.
Fasted triglyceride concentration | Change from baseline fasted triglyceride concentration at 8 weeks.
  A fasted blood sample will be drawn to measure triglyceride concentrations before and after the intervention.
Fasted total cholesterol concentration | Change from baseline fasted total cholesterol concentration at 8 weeks.
  A fasted blood sample will be drawn to measure total cholesterol concentrations before and after the intervention.
Fasted high-density lipoprotein cholesterol concentration | Change from baseline fasted high-density lipoprotein cholesterol concentration at 8 weeks.
  A fasted blood sample will be drawn to measure high-density lipoprotein cholesterol concentrations before and after the intervention.
Fasted low-density lipoprotein cholesterol concentration | Change from baseline fasted low-density lipoprotein cholesterol concentration at 8 weeks.
  A fasted blood sample will be drawn to measure low-density lipoprotein cholesterol concentrations before and after the intervention.
Fasted C-reactive protein concentration | Change from baseline fasted C-reactive protein concentration at 8 weeks.
  A fasted blood sample will be drawn to measure C-reactive protein concentrations before and after the intervention.
Fasted insulin concentration | Change from baseline fasted insulin concentration at 8 weeks.
  A fasted blood sample will be drawn to measure insulin concentrations before and after the intervention.
Fasted glucose concentration | Change from baseline fasted glucose concentration at 8 weeks.
  A fasted blood sample will be drawn to measure glucose concentrations before and after the intervention.
Arterial stiffness | Change from baseline arterial stiffness at 8 weeks.
  Aortic pulse wave velocity will be used to assess arterial stiffness, an independent predictor of cardiovascular disease risk. A noninvasive device (Vicorder) will be used to assess arterial stiffness which measures pulse wave velocity between the carotid and the femoral arteries.
QRISK2 questionnaire | Change from baseline QRISK2 questionnaire at 8 weeks.
  QRISK2 is a cardiovascular disease (CVD) risk score which is designed to estimate the risk of a person developing CVD over the next 10 years. This will be assessed using a short questionnaire before and after the intervention.
Weight | Change from baseline weight at 8 weeks.
  Weight in kilograms will be measured using an electronic measuring station before and after the intervention.
Body mass index | Change from baseline body mass index at 8 weeks.
  Height in cm and weight in kilograms will be measured and combined to calculate body mass index in kg/m^2 before and after the intervention.
Medical Research Council dyspnoea scale | Change from baseline MRC dyspnoea scale at 8 weeks.
  The Medical Research Council dyspnoea scale is a questionnaire that assesses how breathlessness affects COPD patient mobility. The questionnaire will be completed before and after the intervention. The scale range from 1 to 5. as 5 is the worse.
Borg Breathlessness score | Change from baseline Borg breathlessness score at 8 weeks.
  The Borg breathlessness scale is a questionnaire that assesses pateint breathlessness. The questionnaire will be completed before and after the intervention. The scale range is from 0 to 10 as 0 no difficulty in breathing and 10 is the maximum breathlessness score.
Step counts per day | Change from baseline step counts per day at 8 weeks.
  Physical activity level (step count per day) will be measured using an actigraph physical activity monitor. Participants will wear the device for one week on two occasions at week 1 (before the intervention) and week 8 (after the intervention).
Chronic Respiratory Disease Questionnaire Self-Reported(CRQ-SR) | Change from baseline CRQ-SR at 8 weeks.
  CRQ-SR is used to measure the health status of COPD patients. The questionnaire will be completed before and after the intervention.
Bristol COPD Knowledge Questionnaire (BCKQ) | Change from baseline BCKQ at 8 weeks.
  BCKQ is a questionnaire that is used to assess the knowledge that is appropriate for COPD patients. The questionnaire will be completed before and after the intervention.
COPD Assessment Test (CAT) Questionnaire | Change from baseline CAT at 8 weeks.
  The CAT questionnaire it is designed to measure the impact of COPD on a person's life. The questionnaire will be completed before and after the intervention.
Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS at 8 weeks.
  HADS is a self-rating scale that measures anxiety and depression. The questionnaire will be completed before and after the intervention. The scale score range from 0 to 21. 0-7 considered normal, 8 to 10 is considered borderline abnormal and 11 to 21 is considered abnormal.
Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) | Change from baseline PRAISE at 8 weeks.
  PRAISE is a tool that predicts the reduction in sedentary time following pulmonary rehabilitation in individuals with chronic obstructive pulmonary disease (COPD). UIt will be completed before and after the intervention.
The Incremental Shuttle Walking Test (ISWT) | Change from baseline exercise capacity at 8 weeks.
  The Incremental Shuttle Walking Test (ISWT) in meters will be completed before and after the intervention to assess exercise capacity.
The endurance shuttle walk test (ESWT) | Change from baseline exercise capacity at 8 weeks.
  The endurance shuttle walk test (ESWT) in minutes will be completed before and after the intervention to assess exercise capacity.

SECONDARY OUTCOMES:
Postprandial triglyceride concentrations (sub-group only) | Change from baseline postprandial triglyceride concentration at 8 weeks.
  Triglyceride concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial TAG response. The test will be conducted before and after the intervention.
Postprandial total cholesterol concentration (sub-group only) | Change from baseline postprandial total cholesterol concentration at 8 weeks.
  Total cholesterol concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial total cholesterol response. The test will be conducted before and after the intervention.
Postprandial high-density lipoprotein cholesterol concentration (sub-group only) | Change from baseline postprandial high-density lipoprotein concentration level at 8 weeks.
  High-density lipoprotein cholesterol concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial high-density lipoprotein cholesterol response. The test will be conducted before and after the intervention.
Postprandial low-density lipoprotein cholesterol concentration (sub-group only) | Change from baseline postprandial low-density lipoprotein cholesterol concentration at 8 weeks.
  Low density lipoprotein cholesterol concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial low density lipoprotein cholesterol response. The test will be conducted before and after the intervention.
Postprandial total C-reactive protein concentration (sub-group only) | Change from baseline postprandial C-reactive protein concentration at 8 weeks.
  C-reactive protein concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial C-reactive protein response. The test will be conducted before and after the intervention.
Postprandial total insulin concentration (sub-group only) | Change from baseline postprandial insulin concentration at 8 weeks.
  insulin concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial insulin response. The test will be conducted before and after the intervention.
Postprandial total glucose concentration (sub-group only) | Change from baseline postprandial glucose concentration at 8 weeks.
  Glucose concentrations will be measured after an overnight fast and 4 h after consuming a high-fat meal to measure the postprandial glucose response. The test will be conducted before and after the intervention.
Visceral adipose tissue | Baseline visceral adipose tissue
  Visceral adipose tissue will be quantified before the intervention using magnetic resonance imaging (MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Sally Singh, Professor, Study Chair — University Hospital of Leicester NHS Tust
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Siegrist J. Physical activity and risk of cardiovascular disease--a meta-analysis of prospective cohort studies. Int J Environ Res Public Health. 2012 Feb;9(2):391-407. doi: 10.3390/ijerph9020391. Epub 2012 Jan 26. PMID 22470299
- [Background] Gimeno-Santos E, Frei A, Steurer-Stey C, de Batlle J, Rabinovich RA, Raste Y, Hopkinson NS, Polkey MI, van Remoortel H, Troosters T, Kulich K, Karlsson N, Puhan MA, Garcia-Aymerich J; PROactive consortium. Determinants and outcomes of physical activity in patients with COPD: a systematic review. Thorax. 2014 Aug;69(8):731-9. doi: 10.1136/thoraxjnl-2013-204763. Epub 2014 Feb 20. PMID 24558112
- [Background] Triest FJ, Singh SJ, Vanfleteren LE. Cardiovascular risk, chronic obstructive pulmonary disease and pulmonary rehabilitation: Can we learn from cardiac rehabilitation? Chron Respir Dis. 2016 Aug;13(3):286-94. doi: 10.1177/1479972316642367. Epub 2016 Apr 14. PMID 27081189
- [Background] Shortreed SM, Peeters A, Forbes AB. Estimating the effect of long-term physical activity on cardiovascular disease and mortality: evidence from the Framingham Heart Study. Heart. 2013 May;99(9):649-54. doi: 10.1136/heartjnl-2012-303461. Epub 2013 Mar 8. PMID 23474622
- See also: Global Initiative for Chronic Obstructive Lung Disease (GOLD). Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD). . 2017 — http://goldcopd.org